CLINICAL TRIAL: NCT02446340
Title: A Double-Blind, Placebo-Controlled Multiple Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of ShK-186
Brief Title: Multiple Ascending Dose Safety Study of ShK-186 (Dalazatide) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kineta Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 186-02
Record Dates: First submitted 2015-04-15; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: ShK-186; dalazatide; Kv1.3; SHK
MeSH Terms: interventions — Shk-186 peptide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- dalazatide 5ug (Experimental): 8 subjects, 6 given active agent and 2 given placebo
  Interventions: Drug: dalazatide; Drug: placebo
- dalazatide 15ug (Experimental): 8 subjects, 6 given active agent and 2 given placebo
  Interventions: Drug: dalazatide; Drug: placebo
- dalazatide 30ug (Experimental): 8 subjects, 6 given active agent and 2 given placebo
  Interventions: Drug: dalazatide; Drug: placebo
- dalazatide 60ug (Experimental): 8 subjects, 6 given active agent and 2 given placebo
  Interventions: Drug: dalazatide; Drug: placebo

INTERVENTIONS:
Drug: dalazatide — Different doses of drug, subcutaneous injection twice per week for a total of 9 doses.
  Other Names: ShK-186
Drug: placebo — Placebo delivered via subcutaneous administration twice per week for a total of 9 doses
  Other Names: Sub Q Placebo

SUMMARY:
The purpose of this study is to examine safety outcomes in healthy volunteers after systemic administration of multiple ascending doses of dalazatide.

DETAILED DESCRIPTION:
The purpose of this study is to examine safety outcomes in healthy volunteers after systemic administration of multiple ascending doses of dalazatide delivered via subcutaneous injection twice per week for a total of 9 doses.

ELIGIBILITY:
Inclusion Criteria:

1. healthy normal male and female subjects, ages 18 to 45, inclusive;
2. able to communicate and able to provide valid, written informed consent;
3. within the body mass index (BMI) range of approximately 18.0 to 30.0 kg/m2, inclusive;
4. minimum weight of 50 kg;
5. willingness to remain totally abstinent or use adequate contraception; e.g., 2 of the following methods: hormonal contraceptive, intrauterine device, condom, diaphragm, and spermicidal gel/foam) in order to prevent pregnancy from the screening visit until 60 days after the follow-up visit. For men, the donation of sperm during this period is also prohibited.

Exclusion Criteria:

1. the presence of clinically significant medical history as determined by the investigator.
2. the history of clinically significant cardiac abnormalities or presence of clinically significant abnormality on 12-lead ECG.
3. the history of pre-existing paresthesia or neuropathy;
4. abnormalities on neurologic exam at screening or baseline
5. the history of any cancer requiring systemic chemotherapy or radiation; individuals with a history of non-melanoma skin cancer, nonrecurring carcinoma in situ treated with laser or cryotherapy or cervical cancer-in-situ, resected surgically with no evidence of disease, may be accepted on a case by case basis at the discretion of the Investigator;
6. the presence of acute infection or history of acute infection within 7 days prior to receipt of the study drug; additionally, oral temperature may not exceed 37.4°C at baseline;
7. the presence of clinically significant laboratory abnormalities (chemistry panel of 20 analytes [Chem-20; fasted 10-12 hours], complete blood count [CBC], and urinalysis [UA]) as determined by the investigator;
8. positive urine drug screen for drugs of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines, cotinine, tricyclic antidepressants and alcohol) at Screening or at Baseline.
9. typical intake of more than 7 units of alcohol per week (one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
10. a positive hepatitis screen (Hepatitis BsAg or anti-HCV) or positive Human Immunodeficiency Virus (HIV) antibody test ;
11. a history of multiple drug allergies that are important in the view of the Investigator;
12. any history of anaphylaxis or a history of allergy to a medication, diet, or environmental exposure (including bee stings) that are important in the view of the Investigator;
13. participation in another clinical trial with receipt of an investigational product within 60 days of dose administration (or 5 half lives, whichever is longer);
14. recent (within 1 year of Screening) history of illicit drug use;
15. history of alcohol abuse that is important in the view of the Investigator
16. inadequate venous access that would interfere with obtaining blood samples;
17. use of prescription medications, over the counter products, herbal remedies and nutritional supplements within 7 days of study drug administration and throughout the study, or the anticipated need for prescription medications prior to Study Completion;
18. recipients of blood transfusion or transfusion of blood or plasma products within 60 days of study drug administration;
19. donation of blood > 500 mL within 2 months of study drug administration;
20. positive pregnancy test at screening or at baseline (female subjects only);
21. history within the past 3 months of eating disorders or other conditions which may lead to suspicion about the participant's nutritional status;
22. inability or unwillingness to comply with study restrictions

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Subjects with adverse events | From randomization to Day 57 (14 time points)

SECONDARY OUTCOMES:
Subjects with changes in vital signs | From randomization through Day 57 (14 time points)
  Vital signs include temperature, respiratory rate, supine blood pressure and pulse.
Subjects with changes in symptom-directed physical examinations | From date of randomization to day 57 (14 timepoints)
Subjects with changes in 12-lead electrocardiograms | From date of randomization to day 57 (5 timepoints)
PK parameters | pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 4 hours post dose, 8 hours post dose, 12 hours post dose
  Parameters include Area under the plasma concentration versus time curve of dalazatide (AUC)
Presence of specific anti-drug antibody | From date of randomization through Day 57 (4 timepoints).
  Serum evaluated for specific anti-drug antibody using ELISA-based immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Iadonato, PhD, Study Chair — Kineta Inc.
Locations (1):
- PRA International, Lenexa, Kansas, United States